CLINICAL TRIAL: NCT03965624
Title: A Prospective Open-label Trial to Assess the Efficacy and Safety of Ixazomib and Dexamethasone in Patients With Refractory Autoimmune Cytopenia
Brief Title: Efficacy and Safety of Ixazomib and Dexamethasone Refractory Autoimmune Cytopenia
Acronym: Ixa-Cyto
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision of sponsor: impossibility of contract with Takeda
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Takeda Pharmaceuticals International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P171201J; 2018-004556-38 (EudraCT Number)
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2018-12

CONDITIONS: Immune Thrombocytopenia; Warm Autoimmune Hemolytic Anemia
Keywords: MCNS; Rituximab; Complete remission
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Pathologic Complete Response | interventions — ixazomib

STUDY DESIGN:
Intervention Model Description: Prospective interventional uncontrolled single arm open study evaluating the rate of patients achieving 5 cycles without severe toxicity and response on therapy: Interventional clinical study phase IIb , Non-comparative, Not randomised, Not controlled, Unblinded.
  Oral ixazomib will be given on days 1, 8, 15 of a 28-days cycle, in combination with dexamethasone 20 mg weekly. The investigator will start with first test dose levels of ixazomib of 3 mg and process with dose escalation, in case of non-response and no severe adverse events at cycle 1 or de-escalation in case of response and severe adverse events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ixazomib (Experimental): Oral ixazomib will be given on days 1, 8, 15 of a 28-day cycle, in combination with dexamethasone 20 mg weekly. The investigator will start with first test dose levels of ixazomib of 3 mg and process with dose escalation, in case of non-response and no severe adverse events at cycle 1 (see below) or de-escalation in case of response and severe adverse events.
  Interventions: Drug: Ninlaro

INTERVENTIONS:
Drug: Ninlaro — Oral ixazomib will be given on days 1, 8, 15 of a 28-day cycle, the investigator will start with first test dose levels of ixazomib of 3 mg and process with dose escalation, in case of non-response and no severe adverse events at cycle 1 (see above) or de-escalation in case of response and severe adverse events.
  Other Names: Ixazomib

SUMMARY:
Some patients with antibody-mediated autoimmune hematological diseases (warm autoimmune hemolytic anemia (wAIHA), cold agglutinin disease (cAIHA) and immune thrombocytopenia (ITP)) shows no or only minor and transient response to therapy despite several treatment-lines. Such patients are more likely to have a severe disease, with a higher morbidity and mortality.

Hypothesis Effective depletion of autoreactive plasma cells might be the key for a curative approach of these diseases. Therefore, there is a rationale for using proteasome inhibitors (PIs) in these refractory patients.

The rationale is that non-tumoral autoreactive plasma cells are rapidly targeted by proteasome inhibitors. It led us to propose a short course of dexamethasone and ixazomib (5 cycles), to evaluate the safety/efficacy of this innovative strategy of treatment.

Method Prospective interventional uncontrolled single arm open study evaluating the rate of patients achieving 5 cycles of ixazomib and dexamethasone without severe toxicity and response on therapy.

ELIGIBILITY:
Inclusion Criteria:

ITP patients:

1. Age >= 18 years
2. Diagnosis of ITP according to the international definition (Rodeghiero et al Blood 2009)
3. Platelets count < 30 x 109/L or <50 x 109/L if presence of hemorrhagic events or other reason left up to investigator discretion within the months preceding inclusion.
4. Multirefractory ITP defined as patients who have previously failed to maintain a response after rituximab (anti-CD20), splenectomy, and romiplostim and eltrombopag, except if patients have any contraindications or refused these treatments

wAIHA patients

1. Age >= 18 years
2. Diagnosis of wAIHA , symptomatic anemia and a positive direct antiglobulin test
3. Refractory AIHA who have previously failed to maintain a sustained response after rituximab (anti-CD20) and splenectomy except if patients have any contraindications or refused these treatments.

For all patients;

1. Absolute neutrophil count (ANC) >=1,000/mm3
2. Gammablobulin level > 7 g/l
3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3x ULN.
4. Calculated creatinine clearance >=30 mL/min
5. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion criteria

1. Major surgery within 14 days before enrollment.
2. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
3. Female patients who are lactating or have a positive serum pregnancy test during the screening period.
4. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
5. Systemic treatment, within 14 days before the first dose of ixazomib, with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital, azathioprine), or use of St. John's wort.
6. ) Positive HIV test and/or hepatitis virus C infection and/or positive hepatitis B virus surface antigen or core antibody (HbsAg or HBcAb) and/or Active Varicella or Herpes and zoster infection.
7. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
8. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
9. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing.
10. Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
11. Unable to comply with study and follow-up procedures due to psychiatric disorders or any other reason.
12. Inflammatory central nervous system disorder.
13. Patient has >=Grade 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period.
14. Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.
15. Patients that have previously been treated with ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not.
16. Total bilirubin ≥ 1.5 x the upper limit of the normal range (ULN).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patients achieving a response (CR+R) with 5 cycles without severe toxicity (grade III/IV) | 6 months
  Criteria of response:
  ITP: A complete response is defined by a platelet count > 100 x 109/L maintained in the absence of any other ITP directed therapies. A responder to treatment is defined by a patient with a maintained platelet count at > 30 x109/L (Rodeghiero et al Blood 2008) and a minimum twofold increase from initial platelet levels in the absence of bleeding and/or use of ITP directed therapies.
  AIHA: Complete response (CR) is defined as normalization in haemoglobin concentration (Hb≥12 g/dL) without any ongoing immunosuppressive treatment and without any biochemical signs of hemolytic activity. Response (R) is defined as a haemoglobin concentration ≥10 g/dL and requiring continued low-dose prednisolone (<20 mg/day prednisone) or at least 2 g/dL increase in Hb, and no transfusion requirement

SECONDARY OUTCOMES:
Number of patients responding to treatment (CR+R) | At Day 28, Day 56, Day 84, Day 112, 6 months, 9 months and 12 months.
  CR=complete response, R= Response
Number of patients experiencing a A treatment-emergent adverse event (TEAE) along the course of the study. | Up to 12 months
  A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug (AE start date ≥ first dose date) and within 30 days after receiving the last dose of study drug. TEAE will be scaled according to Common Terminology Criteria for Adverse Events (CTCAE) version 4. A severe toxicity severe toxicity is defined as ≥ grade III.
  For ITP patients, thrombocytopenia will not be included in TEAE if it is due to disease activity. But severe bleeding manifestations as unexpected severe hemorrhagic events defined as intracranial hemorrhage, gastrointestinal or visceral bleeding with a decrease of hemoglobin by more than 2 g/dl should be reported as SAE.
  For AIHA patients, anemia will not be included in TEAE if it is due to disease activity. But, severe, unexpected anemia (less thant 6 g/dl) in patients who have previously achieved a response should be reported as SAE.
Gammablobulin level (and isotype) along the study | Day 28, Day 56, Day 84, Day 112, 9 months and 12 months
Number of infectious events along the study | Up to 12 months
Number of bleeding manifestations according to the French bleeding score for ITP patients | At Day 28, Day 56, Day 84, Day 112, 6 months, 9 months and 12 months.
Protective antibody titers (measles, mumps, tetanus) (Ancillary Study) | Day 0, Day 84, 6 months, 9 months and 12 months
Number of pathogenic circulating plasmablasts (Ancillary study) | Day 0, 28, 56, 84, 112 months 6, 9, 12 months
Number and program of bone marrow pathogenic plasma cells for patients with refractory disease (Ancillary study). | Day 0, 6 months
Anti-platelets/red blood cells antibodies (Ancillary study) | Day 0, Day 84, 6 months
Level of serum cytokines (Ancillary study) | Day 0, Day 28, Day 56, Day 84, Day 112 and 6 months , 9 months , 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Mahevas, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Mahevas, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION